CLINICAL TRIAL: NCT02037074
Title: A Double-Blind, Escalating Dose Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Evaluation of Repeat Doses of EVP-6308 or Placebo in Subjects With Schizophrenia on a Stable Antipsychotic Regimen
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetic (PK) and Pharmacodynamic (PD) Effects of EVP-6308 and the Potential of EVP-6308 to Affect the PK Properties of the Antipsychotic Regimen in Subjects With Schizophrenia Currently Receiving Stable Treatment With up to 2 Atypical Antipsychotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-6308-003
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Schizophrenia
Keywords: Phosphodiesterase 10 inhibitor
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Experimental: EVP-6308; Arm 1 (Experimental): low dose, Capsule, Twice Daily, Day 1 through Day 14
  Interventions: Drug: Drug: EVP-6308
- Experimental: EVP-6308; Arm 2 (Experimental): intermediate dose, Capsule, Once Daily, Day 1 through Day 14
  Interventions: Drug: Drug: EVP-6308
- Experimental: EVP-6308; Arm 3 (Experimental): high dose, Capsule, Once Daily, Day 1 through Day 14
  Interventions: Drug: Drug: EVP-6308
- Placebo Comparator; Arm 4 (Placebo Comparator): Placebo, Capsule, Once Daily, Day 1 through Day 14
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug: EVP-6308 — Arms 1, 2, 3
  Arms: Experimental: EVP-6308; Arm 1; Experimental: EVP-6308; Arm 2; Experimental: EVP-6308; Arm 3
Drug: Placebo — Arm 4
  Arms: Placebo Comparator; Arm 4

SUMMARY:
This is a randomized, double-blind, placebo-controlled, sequential cohort, ascending oral dose study of the safety, tolerability, pharmacokinetics, and pharmacodynamics of EVP-6308 administered for 14 days in subjects with schizophrenia who are on a stable anti-psychotic regimen.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosed with schizophrenia, male or female subjects, 18 to 60 years of age

Exclusion Criteria:

* Clinically significant abnormalities on physical examination, medical history, ECG, vital signs, laboratory values, or unstable medical or psychiatric illness
* Any disorder that may interfere with drug absorption
* Clinically significant allergy or sensitivity to medications Positive test for human immunodeficiency virus (HIV) antibodies, Hepatitis B surface antigen, or Hepatitis C antibody
* Pregnant or breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of EVP-6308 in subjects with schizophrenia currently receiving stable treatment with up to 2 atypical antipsychotics | Baseline to Day 21 or Early Termination
  Vital signs measurements, Clinical laboratory tests, Physical examination, ECG findings, Columbia-Suicide Severity Rating Scale. Adverse events and concomitant medications will be collected from the time of signing the informed consent.

SECONDARY OUTCOMES:
Pharmacokinetics of EVP-6308 in subjects with schizophrenia and the potential for EVP-6308 to affect the pharmacokinetic properties of the antipsychotic regimen | Day -1 through Day 16
  PK parameters to be determined for EVP-6308 and EVP-6308 N-oxide metabolite include Cmax, Tmax,, AUC, and t1/2. PK parameters to be determined for the antipsychotic include Cmax, Tmax, AUC, and CL/F.
Potential pharmacodynamics effects of EVP-6308 | Baseline to Day 21 or Early Termination
  Quantitative EEG, Positive and Negative Syndrome Scale, Clinician Global Impression - Severity, Barnes Akathisia Rating Scale, Simpson-Angus Scale, Abnormal Involuntary Movement Scale, Cognitive Battery.

CONTACTS AND LOCATIONS:
Locations (1):
- Long Beach, California, United States